CLINICAL TRIAL: NCT01821183
Title: Strength and Strength-ratio of Hip Rotator Muscles at Soccer Players Compared to Non-soccer Players
Brief Title: Strength and Strength-ratio of Hip Rotator Muscles at Soccer Players
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: c.b.1.1
Record Dates: First submitted 2013-03-26; First posted 2013-03-29 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Hip Injuries; Muscular Atrophy; Dysfunction
MeSH Terms: conditions — Hip Injuries; Muscular Atrophy

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- hip rotators muscle strength
- control group: no intervention

SUMMARY:
At this investigation we want to find out whether there is a difference in muscle strength of the internal and external rotation hip muscles between soccer players and non-soccer players caused by typical movement patterns seen in soccer sport.

DETAILED DESCRIPTION:
Nontraumatic hip injuries are a problem often seen in Soccer Players. A biomechanical formation mechanism is probably. Little research has focused on the measurement of hip external and internal rotation strength at soccer players. The purpose of this study is to investigate the influence of soccer sports at the isometric force and force ratio of the hip rotator muscle system. Two samples of Athletes will be compared: Soccer Players (N15) and Non-soccer players (N15) matched in sex, age and level of physical activity to investigate hip rotator force in 3 different angles of hip flexion (0°/45°/90°). The measurement will be made with a handheld dynamometer.

ELIGIBILITY:
Inclusion criteria:

Study group:

Amateur footballers (N15) in the age between 18 and 35 At least five years of active footballer's career Football training twice weekly Active participation in play No pain or limitations in the area of the hip or the lower extremity

Control group:

Athletes (N15), non-soccer players with now asymmetric leg activities In the age between 18 and 35 At least twice weekly sports activity for at least 30 minutes No pain or limitations in the area of the hip or the lower extremity

Exclusion criteria:

Professions with asymmetric leg activities Pain or limitations in the area of the hip or the lower extremity Surgery on the hip in the prehistory

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: soccer club of Sarnen, Switzerland Residents of Sarnen and Basel, Switzerland
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Strength of the internal and external rotators of the hip | "up to 10 months"

CONTACTS AND LOCATIONS:
Overall Officials: Niklaus F. Friederich, MD Professor, Principal Investigator — Head of degree program: Master of Functional Kinetic Science, University of Basel, Switzerland
Locations (1):
- Physiotherapy Burch&Keiser, Sarnen, Canton of Obwalden, Switzerland